CLINICAL TRIAL: NCT02632565
Title: Intra-Articular 0.5 % Lidocaine Injection Under Ultrasound Guidance in Chronic Knee Pain Due To Osteoarthritis
Brief Title: Intra-Articular 0.5 % Lidocaine Injection for Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: H. Evren Eker (Other)
Collaborators: Baskent University (Other)
Responsible Party: Sponsor-Investigator, H. Evren Eker, Ass Prof, Baskent University
Organization: Baskent University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KA08/83
Record Dates: First submitted 2015-12-03; First posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Pain
Keywords: osteoarthritis; lidocaine; pain; ultrasound
MeSH Terms: conditions — Chronic Pain; Osteoarthritis; Pain | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intra-articular 0.5% lidocaine (Active Comparator): intra-articular 7 mL 0.5% lidocaine injection for 3 times with one week intervals
  Interventions: Drug: Lidocaine
- intra-articular saline (Active Comparator): intra-articular 7 mL saline injection for 3 times with one week intervals
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Lidocaine
  Arms: intra-articular 0.5% lidocaine
Drug: Saline
  Arms: intra-articular saline

SUMMARY:
In this study, investigators compared the efficacy of intra-articular 0.5% lidocaine and saline injection on pain, stiffness and physical function in patients with osteoarthritis.

DETAILED DESCRIPTION:
Patients with osteoarthritis were randomly allocated into two groups. Group I (n=26) received intra-articular injection of 7 mL 0.5% lidocaine and Group II (n=26) received 7 mL saline into painful knee for 3 times with one week intervals under USG guidance. VAS and WOMAC scale including pain, stiffness and physical function was used for the assessment of patients with osteoarthritis. Analgesic requirements were also recorded.

The primary outcome parameter of this study was the pain scores. The sample size for the primary variable was calculated based on a standard deviation of 20 mm estimated from a previous study. A power analysis with a type II error of 20% at a two-sided 5% significance level estimated 22 patients per group to be included. Investigators included 26 patients per groups for possible missing date. χ2 test for categorical data and independent samples t-test for the comparison of VAS and WOMAC scores between groups were used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* knee pain for more than 25 of the past 30 days, morning stiffness or less than 30 minutes, crepitation in the knee
* pain for more than 25 of the past 30 days and osteophytes on x-ray examination of the knees indicating knee OA

Exclusion Criteria:

* the knees with a history of mechanical derangement, fibromyalgia, skin lesions and other risk factors of infection, therapy with anticoagulants and trauma/surgery

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-12; Primary Completion 2015-03 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Pain scores according to visual analog scale | 3 months after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anis Aribogan, Prof, Study Chair — Coordinator

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elhakim M, Nafie M, Eid A, Hassin M. Combination of intra-articular tenoxicam, lidocaine, and pethidine for outpatient knee arthroscopy. Acta Anaesthesiol Scand. 1999 Sep;43(8):803-8. doi: 10.1034/j.1399-6576.1999.430804.x. PMID 10492407
- [Background] Pietruck C, Grond S, Xie GX, Palmer PP. Local anesthetics differentially inhibit sympathetic neuron-mediated and C fiber-mediated synovial neurogenic plasma extravasation. Anesth Analg. 2003 May;96(5):1397-1402. doi: 10.1213/01.ANE.0000060454.34258.D3. PMID 12707141